CLINICAL TRIAL: NCT03120871
Title: Sex Differences in Youth-Onset Type 2 Diabetes: Exploring Mechanisms
Brief Title: Microbiome Insulin Sensitivity Study
Acronym: MISS
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Children's Hospital Colorado (Other)
Responsible Party: Sponsor
Other Study IDs: 16-2633; UL1TR001082 (NIH)
Record Dates: First submitted 2017-04-14; First posted 2017-04-19 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Obesity; Insulin Resistance; Type2 Diabetes
Keywords: Beta cell failure; Puberty; Microbiome; Insulin Sensitivity
MeSH Terms: conditions — Obesity; Insulin Resistance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Stool, urine, and serum and plasma will be collected and banked for future research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All subjects: Female sex, obese, aged 9-17 years, Tanner stages 1-5.

SUMMARY:
The Microbiome Insulin Sensitivity Study "MISS" is a pilot study designed to study microbiome composition across puberty and how it relates to insulin sensitivity and secretion in obese girls, who are at increased risk for developing type 2 diabetes in puberty. The investigators will evaluate the gut microbiome composition in fecal samples of 57 obese girls in three groups: prepubertal (Tanner 1), early pubertal (Tanner 2-3), and late pubertal (Tanner 4-5). Insulin sensitivity will also be measured via an intravenous glucose tolerance test (IVGTT) in 18 prepubertal and late pubertal participants.

DETAILED DESCRIPTION:
Pediatric type 2 diabetes (T2D) is increasing in prevalence and its incidence is twice as high in girls as in boys. Pediatric onset of T2D occurs exclusively in obese youth and is tightly linked with puberty, suggesting a link with the physiologic insulin resistance of puberty. However, markers are as yet unavailable to identify those at highest risk for progression to T2D. Results from the Treatment Options for Diabetes in Youth (TODAY) Study demonstrate that pediatric T2D appears to progress rapidly in youth, forecasting poor quality of life and early complications. Therefore, identifying those most at risk and developing a better understanding of the pathophysiology of onset of T2D in youth are critical for preventing T2D, particularly in obese girls.

The investigators overarching hypothesis is that effects of obesity on metabolic and hormonal changes during puberty place obese girls at greatest risk for early T2D, similar to that which is seen in women with gestational diabetes. More specifically, sex steroid effects on insulin resistance, β-cell function, and body composition may contribute to both the pubertal increase in risk for T2D, as well as the disproportionately higher prevalence of T2D among girls. The investigators long-term goal is to design a focused intervention aimed to prevent progression to T2D during puberty. In order to do this it is necessary to: 1. Develop a better understanding of underlying mechanisms for β-cell failure in obese youth during puberty, and 2. Identify early markers for predicting which obese youth will progress to early T2D.

Alterations in gut microbiota appear to play an important role in mediating obesity and insulin resistance through poorly understood mechanisms. Current hypotheses are that shifts in the composition of the gut microbiome lead to dysregulation of complex polysaccharide metabolism, altered production of gut hormones regulating energy balance, and local and systemic inflammation. The gut microbiome composition has been reported to change during pregnancy and may play a role in metabolic changes during this time. As metabolic and hormonal changes in puberty parallel those in pregnancy, shifts in the microbiome may also accompany metabolic shifts during puberty. Currently, there are no published studies evaluating shifts in human gut microbiome composition during puberty. Consequently, the overall goal of this study is to collect cross-sectional preliminary data to inform feasibility of a future longitudinal study of metabolic and hormonal changes in lean and obese youth during the pubertal transition.

ELIGIBILITY:
Inclusion Criteria:

* Female sex
* Obesity (BMI > 95th percentile for age)
* Age > 9 years, <18 years

Exclusion Criteria:

* Medications affecting glucose metabolism
* Known T2D
* Known polycystic ovarian syndrome
* Known fatty liver disease (ALT > 2x above the upper limit of normal)
* Chronic illness affecting glucose metabolism
* Antibiotic use in the previous 6 months

Ages: 9 Years to 17 Years | Sex: Female
Age Groups: Child
Gender Based: Yes — Participants must be biologically female
Study Population: 19 prepubertal (Tanner 1, [T1]), 19 early pubertal (T2-3), 19 late pubertal (T4-5) obese (BMI>95%ile) females, age >9 years.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2018-08-19 (Actual); Study Completion 2018-08-19 (Actual)

PRIMARY OUTCOMES:
Firmicutes:Bacteroides ratio (F:B Ratio) | Within 2 weeks of enrollment
  F:B ratio in prepubertal, early pubertal, and late pubertal obese girls by high-throughput 16S ribosomal ribonucleic acid (16 S rRNA) sequencing from stool samples.
Insulin sensitivity (Si) | Within 2 weeks of enrollment
  Insulin sensitivity (Si) estimated from IV glucose tolerance testing using Bergman's minimal model

SECONDARY OUTCOMES:
Urinary estradiol metabolites (E1c) | Within 2 weeks of enrollment
  Measurement of estrogen metabolites in first morning urine sample and normalized to creatinine
Urinary luteinizing hormone (LH) | Within 2 weeks of enrollment
  Measurement of LH in first morning urine sample and normalized to creatinine
Urinary follicle stimulating hormone (FSH) | Within 2 weeks of enrollment
  Measurement of FSH in first morning urine sample and normalized to creatinine

CONTACTS AND LOCATIONS:
Overall Officials: Megan M Kelsey, MD, MS, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No